CLINICAL TRIAL: NCT04090593
Title: Chronic Disease Mobile Educational Experience for Hospitalized Patients
Brief Title: Chronic Disease Mobile Educational Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS-19-00145
Record Dates: First submitted 2019-08-13; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Chronic Disease; Heart Failure
MeSH Terms: conditions — Chronic Disease; Heart Failure

STUDY DESIGN:
Intervention Model Description: Study is randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will determine patient eligibility and recruit participants, team will randomize patients to receive intervention vs. current practice. Outcome assessor(s) will be blinded from patient intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Module Intervention (Experimental): Intervention arm patients receive educational mobile module related to chronic condition that contributed to reason for admission.
  Interventions: Other: Patient Education 101: Mobile Health Education Tool
- Hospital Practice Control (No Intervention): Control arm patients receive current, standard practice as related to patient education in the hospital (this does not include an educational mobile module).

INTERVENTIONS:
Other: Patient Education 101: Mobile Health Education Tool — Intervention is interactive, mobile (tablet-or-smart-phone delivered), educational module that patients engage with during hospital admission.
  Arms: Educational Module Intervention

SUMMARY:
This study evaluates the effectiveness of a mobile health education module, in increasing hospitalized patients' understanding of their chronic illness, and in reducing 30-day hospital readmission rates. Half of the participants will receive the educational module intervention in addition to standard education, the other half will receive hospital standard practice education only.

DETAILED DESCRIPTION:
Chronic disease is the leading cause of death and disability, costing the US healthcare system 1 trillion dollars annually. Successful management of these conditions critically requires patient understanding and engagement. Patients are advised to adhere to medications, redesign lifestyles, and navigate the health care system. Most of these care plan items require careful instruction and confirmation of shared understanding.

Mobile health technology has the potential to assist greatly with patient education, especially for hospitalized patients. This prospective study evaluates a specific mobile technology intervention, an educational and emotionally-engaging video patients watch while admitted for a complication related to one of these chronic diseases: Heart Failure, Diabetes, COPD, Asthma, Cirrhosis, Atrial Fibrillation, Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* admission to medical service primary team for decompensation or complication of chronic disease.(e.g. heart failure)

Exclusion Criteria:

* cognitive disability or visual/auditory limitation that prevents self-interaction with educational module

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
30-Day hospital readmission rate | 9 months (270 days)
  In this study, 30-Day hospital readmission rate is defined as the ratio of patients discharged from LAC+USC Medical Center who are readmitted to either LAC+USC Medical Center or one of three other LA County Department of Health Services (DHS) hospitals. (These are Olive View Medical Center, Rancho Los Amigos Hospital, and Harbor-UCLA Medical Center). This rate can be calculated readily by either of two different means: programmed data extraction from the common electronic health record (there is a Power Insight-Cerner report that does this); or blinded, manual chart review.
Self-reported quality of life: Short Form (36) Health Survey | 9 months (270 days)
  As part of the Medical Outcomes Study (MOS), a multi-year, multi-site study to explain variations in patient outcomes, RAND developed the 36-Item Short Form Health Survey (SF-36). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. Survey is attached to this submission.
Patient understanding of chronic disease: 8-item disease focused survey. | 9 months (270 days)
  This study's authors have developed an 8-item survey, each question with equal rate, designed to measure patients' understanding of several key concepts related to their diagnosis and management. The higher the score, the better the presumed understanding. Survey for heart failure is attached to this submission.
Patient satisfaction with treatment: Client Satisfaction Questionnaire (CSQ-8) | 9 months (270 days)
  The CSQ-8 is an 8-item, easily scored and administered measurement that is designed to measure client satisfaction with services. The items for the CSQ-8 were selected on the basis of ratings by mental health professionals of a number of items that could be related to client satisfaction and by subsequent factor analysis. The CSQ-8 is unidimensional, yielding a homogeneous estimate of general satisfaction with services. The higher the score, the better the presumed patient satisfaction with services. Survey is attached to this submission.

CONTACTS AND LOCATIONS:
Overall Officials: Josh Banerjee, MD, MPH, MS, Principal Investigator — LAC+USC Medical Center

IPD SHARING:
Plan to Share IPD: No